CLINICAL TRIAL: NCT06487182
Title: The Effect of Reiki on the Anxiety Level of Mothers Whose Children Receive Hospital Treatment
Brief Title: The Effect of Reiki on the Anxiety Level of Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Director, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/292
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutic Touch; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki (Experimental): The intervention will be applied to the reiki group in the application hospital room. Reiki therapy will be applied by a practitioner with a Reiki application certificate in the application laboratory for 30 minutes while the participants lie down with their eyes closed. 4 sessions of reiki application will be applied to the intervention group for a week. Reiki application will start , the first anxiety scores will be recorded. Anxiety levels after 4 sessions will be recorded.
  Interventions: Other: reiki
- Placebo reiki (Sham Comparator): Placebo Reiki will be applied to the participants in the group in the application hospital room. The practice will be carried out in the application room for 30 minutes, with the participants sitting with their eyes closed. Reiki life energy will not be transferred to participants in the placebo reiki group. Since the participants' eyes are closed, they will not know that there is a transfer. Placebo Reiki application will be performed in the room 4 times during a week. Placebo application will start and the anxiety scores will be recorded. After 4 sessions, anxiety scores will be recorded.
  Interventions: Other: placebo reiki
- control (No Intervention): Routine hospital procedure will be applied. Anxiety scores will be recorded. After a week anxiety scores will be recorded.

INTERVENTIONS:
Other: reiki — reiki
  Other Names: control group; placebo reiki
  Arms: Reiki
Other: placebo reiki — placebo reiki
  Other Names: control group
  Arms: Placebo reiki

SUMMARY:
The aim of this study is to determine the effect of Reiki applied to mothers whose children were treated in the hospital on the anxiety level.

DETAILED DESCRIPTION:
Hypotheses 01; there was no difference between the anxiety score of the reiki group and the anxiety score of the control group.

The study will be carried out in three different groups. The practice will start with meeting the women whose children were treated in the hospital. After the women are evaluated in terms of eligibility criteria for the research, the women who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Reiki Group The intervention will be applied to the reiki group to be applied in the hospital room. Reiki therapy will be applied by a practitioner with a Reiki application certificate in the application laboratory for 30 minutes while the participants lie down with their eyes closed. 4 sessions of reiki application will be applied to the intervention group for a week. Anxiety level after 4 sessions will be recorded.

Placebo Reiki will be applied to the participants in the group in the application hospital room. The practice will be carried out in the application laboratory for 30 minutes, with the participants sitting with their eyes closed. Reiki life energy will not be transferred to participants in the placebo reiki group. Since the participants' eyes are closed, they will not know that there is a transfer. Placebo Reiki application will be performed in the room 4 times during a week. Placebo application will start, and the first anxiety scores will be recorded. After 4 sessions, anxiety scores will be recorded.

control group; the first anxiety scores will be recorded. After a week later anxiety scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* At least the 3rd day of hospitalization

  * Their child has an acute or chronic disease
  * Able to speak and write Turkish and have no communication problems
  * No psychiatric history and not using medication
  * Not drinking alcohol in the last 24 hours
  * Those who have not received body-mind therapy (yoga, reiki, massage, meditation) in the last six months
  * Mothers who volunteer to participate in the research will be included.

Exclusion Criteria:

Reiki practitioner or who also has an instructor

* Having time and communication problems that cannot answer the questions asked
* Mothers who do not volunteer to participate in the study will not be included in the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
anxiety | immediately before reiki application and immediately after the reiki application]
  The State Anxiety Scale assesses feelings of fear, tension, irritability, and anxiety that increase during stress in response to physical danger and psychological stress. The 20-question test allows individuals to answer within 10 minutes.
  It provides answers on a four-point Likert type scale. STAI, reliability ranging from 0.83 to 0.92 It has sufficient validity and reliability with its coefficients (Vitale 2006).

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye BAL, Ph.D., Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)